CLINICAL TRIAL: NCT00456469
Title: Diagnosis of Active and Latent TB Infection With IFN-y Assays in African Children
Acronym: ALTAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Thrasher Research Fund (Other)
Other Study IDs: 06.49 TF Cuevas
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Tuberculosis
Keywords: TB; latent; infection; Ethiopia
MeSH Terms: conditions — Tuberculosis; Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study based in Southern Ethiopia Purpose - to explore if children in contact with adults with TB have positive acute reactants such as IFN-y and other cytokine responses; if these responses discriminate between high and low risk of disease progression and whether these could be incorporated into improved diagnostic approaches.

DETAILED DESCRIPTION:
The study follows children in contact with TB. Those with positive TST will be offered chemoprophylaxis and all children will be followed for 2 years to describe IFN-y responses over time, identify symptoms of active TB and if these symptoms are associated with IFN-y and other cytokine responses.

Children with suspicion of TB attending health centres will also be investigated using routine diagnostic tests and IFN-y and other cytokines responses to evaluate if the latter could be used in improved diagnostic approaches.

ELIGIBILITY:
Inclusion Criteria:

- Children - 1 to 14 years old in contact with adults with smear positive TB

Or:

- Children with suspicion of TB admitted to the hospital for investigations

Exclusion Criteria:

- Residency > 10 Km from recruitment center

Or:

- Patient severely to undergo diagnostic procedures.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500
Dates: Start 2007-05; Study Completion 2009-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Cuevas, Dr, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Bushullo Major Health Centre, Awasa, Southern Region, Ethiopia

REFERENCES:
- [Derived] Yassin MA, Petrucci R, Garie KT, Harper G, Teshome A, Arbide I, Asnake G, Ahmed HJ, Mammo T, Yesuf K, Cuevas LE. Use of tuberculin skin test, IFN-gamma release assays and IFN-gamma-induced protein-10 to identify children with TB infection. Eur Respir J. 2013 Mar;41(3):644-8. doi: 10.1183/09031936.00012212. Epub 2012 Sep 20. PMID 22997219
- [Derived] Garie KT, Yassin MA, Cuevas LE. Lack of adherence to isoniazid chemoprophylaxis in children in contact with adults with tuberculosis in Southern Ethiopia. PLoS One. 2011;6(11):e26452. doi: 10.1371/journal.pone.0026452. Epub 2011 Nov 1. PMID 22069451
- [Derived] Yassin MA, Petrucci R, Garie KT, Harper G, Arbide I, Aschalew M, Merid Y, Kebede Z, Bawazir AA, Abuamer NM, Cuevas LE. Can interferon-gamma or interferon-gamma-induced-protein-10 differentiate tuberculosis infection and disease in children of high endemic areas? PLoS One. 2011;6(9):e23733. doi: 10.1371/journal.pone.0023733. Epub 2011 Sep 23. PMID 21966356